CLINICAL TRIAL: NCT06858488
Title: A Pilot Study on the Technical Feasibility of an Electrical Impedance Tomography Device for Soft Tissue Injury Following High Energy Extremity Fractures
Brief Title: Bioimpedance for Ortho Trauma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Principal Investigator, Ida Leah Gitajn, Section Chief, Orthopaedics, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY02002529
Record Dates: First submitted 2025-02-12; First posted 2025-03-05 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-02

CONDITIONS: Trauma Injury
Keywords: Orthopedics; Extremity fracture
MeSH Terms: conditions — Accidental Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Extremity fracture (Experimental): High energy closed extremity fractures
  Interventions: Procedure: Extremity Surgery

INTERVENTIONS:
Procedure: Extremity Surgery — Patients 18 years of age or older with high energy closed extremity fractures. Provision of informed consent.

SUMMARY:
Patients with high-energy extremity trauma will undergo imaging with an EIT device in the Emergency Department, Operating Room, Orthopaedic Clinic, and In-patient hospital rooms. The EIT device is an electrical impedance tomography system.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* High energy closed extremity fracture
* Provision of informed consent

Exclusion Criteria:

* Metatarsal fractures
* Injury to both lower extremities precluding contralateral imaging
* Presence of an implanted electronic device (e.g. pacemaker, vagal stimulator, deep brain stimulator) or electrodes or electrical wires.
* Currently pregnant, potentially pregnant, or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of the EIT device | 20 minutes
  The primary objective of this work is to explore whether changes in impedance measurement associated with EIT are associated with soft tissue injury and readiness for surgical intervention. EIT is a technique which introduces a small amount of electrical current into biologic tissue through an array of electrodes and measures the change in signal to generate images related to the physiology of that tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Ida L Gitajn, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No